CLINICAL TRIAL: NCT01451983
Title: Genetic, Biochemical, Behavioral and Neuroimaging Phenotypes of Autism Spectrum Disorders (ASDs)
Brief Title: Genetics, Brain Structure and Thinking Skills in Autism
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Thomas W. Frazier, Ph.D, Autism Research Program Director, The Cleveland Clinic
Other Study IDs: CCF 09-624; UL1RR024989 (NIH)
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Results first posted 2015-01-14 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Autism Spectrum Disorders
Keywords: Autism; PTEN; macrocephaly
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Megalencephaly

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — About 6 tubes of blood or up to 50 ml (3-4 tablespoons) and 30 mL of urine will be collected.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- ASD with PTEN: Individuals with autism spectrum disorder who are also found to have a PTEN mutation.
- ASD no PTEN macrocephaly: Individuals with autism spectrum disorder who do not have a PTEN mutation with a large head circumference.
- ASD no PTEN no macrocephaly: Individuals with autism spectrum disorder who do not have a PTEN mutation without a large head circumference.
- Siblings: Siblings of individuals with autism spectrum disorders.

SUMMARY:
The purpose of this research is to better understand the genetic, biochemical, cognitive and behavioral symptom abnormalities that contribute to autism spectrum disorders. The investigators anticipate recruiting at least 100 participants with autism spectrum disorder and large head size, at least 100 participants with autism spectrum disorder without large head size and at least 40 healthy siblings. Biological parents are expected to be recruited only as genetic changes are identified in individuals with autism spectrum disorders to better understand the nature of these genetic changes. Participants are asked to complete cognitive testing, a blood draw, urine collection and measurement of his/her height, weight and head circumference. Parents or caregivers may be asked to complete a diagnostic evaluation and will complete questionnaires that examine the participant's medical and family history as well as his/her current symptoms, functioning, and quality of life. A brief report simply listing and giving a basic description of any behavioral diagnostic information, autism symptoms, adaptive functioning, and a listing of results from cognitive testing will be provided as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of autism
* Consent from parents or guardians or an adult with or suspected of having an autism spectrum disorder that does not require a legal guardian or an adult who is the healthy sibling of an individual with an autism spectrum disorder.
* Youth ages 2-17 and adults ages 18-50. Youths and adults who are able (some young or severely impaired participants may not be able to provide assent) will be asked to provide assent.
* Families with multiple children who meet the above inclusion criteria will be permitted to have as many children participate as they wish.
* Youth ages 2-17 and adults ages 18-50 who do not have an autism spectrum disorder or are not suspected of having an autism spectrum disorder and who have a sibling with an autism spectrum disorder who has participated in the present study.

Exclusion Criteria:

* Clinically significant medical disease that would prohibit participation in the study procedures.
* Children younger than 2 years old and adults older than 50 years old.

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: We anticipate recruiting 80 participants with autism spectrum disorder and large head size, 80 participants with autism spectrum disorder without large head size and 40 healthy siblings. Biological parents are expected to be recruited only as genetic changes are identified in individuals with autism spectrum disorders to better understand the nature of these genetic changes.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2010-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W Frazier, Ph.D., Principal Investigator — The Cleveland Clinic; Charis Eng, M.D., Ph.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Center for Autism, Cleveland, Ohio, United States

REFERENCES:
- See also: Cleveland Clinic Center for Autism Research Website — http://clevelandclinic.org/autismresearch

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ASD With PTEN | ASD no PTEN Macrocephaly | ASD no PTEN no Macrocephaly | Siblings
Started | 26 | 27 | 61 | 24
Completed | 26 | 27 | 61 | 24
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ASD With PTEN | ASD no PTEN Macrocephaly | ASD no PTEN no Macrocephaly | Siblings | Total
Number analyzed (Participants) | 26 | 27 | 61 | 24 | 138
Age, Continuous [Mean (Full Range); unit: years] | 11.9 [2 to 34] | 13.3 [2 to 38] | 9.0 [2 to 45] | 11.7 [2 to 36] | 11.4 [2 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 8 | 10 | 30
  Male | 18 | 23 | 53 | 14 | 108

OUTCOME MEASURES:

1. Primary Outcome: Total Brain Volume
Time Frame: Baseline
Population: MRI acquisition was performed using Siemens Q4 TIM Trio 3 tesla scanner with standard 12-channel receive-only head coil. An 8-minute whole-brain T1-weighted inversion recovery turboflash (MPRAGE) was acquired. Volumetric measurements were obtained using the software suite Freesurfer. Not all participants received imaging due to age and impairment.
Measure: Mean (Standard Deviation); unit: cubic centimeters
Arm/Group | ASD With PTEN | ASD no PTEN Macrocephaly | ASD no PTEN no Macrocephaly | Siblings
Number analyzed (Participants) | 17 | 16 | 38 | 14
cubic centimeters | 1634.1 (272.6) | 1409.8 (158.6) | 1236.7 (121.3) | 1401.9 (199.2)

ADVERSE EVENTS:
Time Frame: 4 years 3 months from May 2010- August 2014
Arm/Group | ASD With PTEN | ASD no PTEN Macrocephaly | ASD no PTEN no Macrocephaly | Siblings
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27 | 0/61 | 0/24
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Modest PTEN-ASD sample size and difficulty in closely matching each PTEN patient to one or more patients from each comparison group; Lack of comprehensively characterized PHTS patients without ASD is also a limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No